CLINICAL TRIAL: NCT00506506
Title: Randomized Controlled Trial Examining the Effect of N-Acetylcysteine on Serum Creatinine in Patients With Stage 3 Chronic Kidney Disease
Brief Title: Effect of N-Acetylcysteine (NAC) on Creatinine in Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Dr. L. Moist, Lawson Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: R-07-358; 13514
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Chronic Kidney Disease
Keywords: N-acetylcysteine; Chronic kidney disease; eGFR; Cystatin C; proteinuria; Stage 3 chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): N-acetylcysteine 1200 mg twice daily x 48 hours
  Interventions: Drug: N-acetylcysteine
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine 1200 mg twice daily x 48 hours
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
N-acetylcysteine is used to reduce the risk of injury to the kidney after the administration of contrast dye. The mechanism and effectiveness of this intervention is not substantiated in the literature. The investigators hypothesize that serum creatinine will be lower in patients who receive NAC compared to those who receive the placebo but serum cystatin C will not change in patients who receive NAC compared to those who receive the placebo. Also urine creatinine will increase after the administration of NAC compared to before the administration of NAC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an eGFR between 30-60 ml/min calculated using last available creatinine and patient weight.
2. Age > 18
3. No known allergies to or adverse effects from NAC
4. No known scheduled radio-contrast procedures
5. No medications known to affect creatinine secretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
24 hour creatinine clearance, estimated glomerular filtration rate (eGFR), proteinuria and cystatin C

CONTACTS AND LOCATIONS:
Overall Officials: Louise Moist, MD, MSC, Principal Investigator — Schulich School of Medicine and Dentistry, University of Western Ontario
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Moist L, Sontrop JM, Gallo K, Mainra R, Cutler M, Freeman D, House AA. Effect of N-acetylcysteine on serum creatinine and kidney function: results of a randomized controlled trial. Am J Kidney Dis. 2010 Oct;56(4):643-50. doi: 10.1053/j.ajkd.2010.03.028. Epub 2010 Jun 11. PMID 20541301